CLINICAL TRIAL: NCT02897245
Title: An Observational Study for CML Patients Who Discontinued Tyrosine Kinase Inhibitors Intentionally After Achieving a Deep Molecular Response
Brief Title: A Study for Tyrosine Kinase Inhibitors Discontinuation
Acronym: A-STIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Philippe ROUSSELOT, Study coordonnator, Versailles Hospital
Other Study IDs: 12/22_aSTIM
Record Dates: First submitted 2016-08-19; First posted 2016-09-13 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Leukemia
Keywords: Myelogenous; Chronic; BCR-ABL Positive
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with intentionally stop
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Treatment of Chronic Myeloid Leukemia (CML) has been revolutionized by the use of tyrosine kinase inhibitors including imatinib mesylate (Gleevec, Novartis Laboratories). Two other inhibitors of the BCR-ABL kinase are currently on the market in France, nilotinib (Tasigna®, Novartis Laboratories) in the first and second-line treatment and dasatinib (SPRYCEL®, Bristol-Myers Squibb Laboratories) in second line. Achieving a complete molecular response (CMR) in patients with Chronic Myeloid Leukemia (CML) treated with tyrosine kinase inhibitors may be currently regarded as the ultimate level of reduction of residual disease. The pilot Stop Imatinib study has opened the way for a french prospective study of stopping imatinib, the STIM study. The results of the STIM study showed that almost 60% of patients exhibited molecular relapse, most frequently within the first 6 months after discontinuation. The parameters that are statistically associated with the loss of complete molecular response are the Sokal score at diagnosis and the total duration of treatment with imatinib. Criteria to define molecular relapse in treatment free remission patients are not well defined and validated. The aim of the study is to validate the loss of major molecular response as a robust criteria for TKI resumption. The patient's population will be CML patients who are offered to discontinue therapy outside the STIM strial.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Chronic Myelogenous leukemia
* mors than 18 years old
* intentionally stop treatment by tyrosine kinase inhibitor

Exclusion Criteria:

* inclusion in a prospective study
* non intentionally stop (adverse event)
* Stop for disease progression
* Death patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These are patients with chronic myeloid leukemia treated with a tyrosine kinase inhibitor for which an intentional discontinuation was made since 2007 outside the framework of a prospective study
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Survival without loss of molecular response major (RMM BCR-ABL / ABL IS ≤ 0.1%) | 2 years

SECONDARY OUTCOMES:
Treatment free survival molecular evolution in treatment discontinuation | 2 years
Progression free survival | 2 years
Overall survival | 2 years
The rate of deep molecular response after restarting TKIs kinase | 2 years
Withdrawal syndrome | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CH Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rousselot P, Loiseau C, Delord M, Cayuela JM, Spentchian M. Late molecular recurrences in patients with chronic myeloid leukemia experiencing treatment-free remission. Blood Adv. 2020 Jul 14;4(13):3034-3040. doi: 10.1182/bloodadvances.2020001772. PMID 32614963